CLINICAL TRIAL: NCT04478149
Title: A Comprehensive Fall Prevention System for Memory Care: Final Feasibility and Randomized Controlled Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SafelyYou (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 241755
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Waitlist control
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Cameras (Experimental): active cameras in the room
  Interventions: Device: SafelyYou
- Inactive Cameras (Sham Comparator): camera in the room, not activated
  Interventions: Other: Control

INTERVENTIONS:
Device: SafelyYou — technology to detect and prevent falls
  Arms: Active Cameras
Other: Control — technology present but not activated
  Arms: Inactive Cameras

SUMMARY:
This study tests novel technology using computer vision and remote clinical review to reduce falls for residents with dementia in assisted living communities.

ELIGIBILITY:
Inclusion Criteria:

* Living in a participating assisted living facility and suffering from dementia

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-31 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Opt-in rate | through study completion, an average of 1 year
  participants enrolling
Number of falls | through study completion, an average of 1 year
  fall incidents
Number of ER visits | through study completion, an average of 1 year
  fall incidents requiring emergency transportation

IPD SHARING:
Plan to Share IPD: No